CLINICAL TRIAL: NCT00148213
Title: Clinical Evaluation of a New Highly Sensitive Thyroglobulin Assay in Differentiated Thyroid Carcinoma
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: Nichols Institute Diagnostika GmbH, Bad Vilbel, Germany (Unknown)
Other Study IDs: CETAT
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2005-09-07 (Estimated); Status verified 2005-09

CONDITIONS: Thyroid Neoplasms
Keywords: differentiated thyroid carcinoma; thyroglobulin; immunoassay; thyroidectomy; radioiodine therapy
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Human thyroglobulin (Tg) is the most sensitive biochemical marker for recurrence of differentiated cancer (DTC), especially after the complete removal of thyroid tissue through surgery and radioiodine therapy (RIT).

Unfortunately, current assays for measuring Tg in blood samples are not sensitive enough to reliably measure Tg while patients are under thyroid hormone replacement therapy. Instead patients have to withdraw thyroid hormone for several weeks or receive costly injections of recombinant thyroid stimulating hormone (TSH) in order to raise Tg production by thyroid remnant and/or thyroid cancer cells so that it can be measured by current Tg assays. Other patients have antibodies against Tg that interfere in current immunoassays.

The purpose of the study was to characterize a new highly sensitive assay for measuring Tg in the serum in thyroid cancer patients both on thyroid hormone therapy and off therapy in comparison to the normal routine assay already in use at Münster University Hospital.

DETAILED DESCRIPTION:
Sera of 100 consecutive DTC patients after total thyroidectomy were to be collected at the Department of Nuclear Medicine both under TSH-suppression therapy and under endogenous TSH stimulation (TSH > 25 mU/l). All patients were staged by clinical examination, cervical ultrasound (7.5 MHz), I-131 whole-body scintigraphy and - where applicable - F18-FDG-PET. Written informed consent was obtained from all pts. Sera were taken in separation tubes without anticoagulants and stored at -20°C until analysis. Sera were allowed to come to room temperature prior to analysis.

Tg, TgR and TgAb concentrations were determined by fully automated two-site chemiluminescence immunoassays (CLIA; Nichols Advantage®; Nichols Institute Diagnostics, San Clemente, California). All 3 assays are based on the identical highly purified hTg material for calibration (Tg), recovery (TgR) and antigen (TgAb; biotinylated and acridinium ester labeled) for optimum comparability of test results.

In addition, Tg and TgR was measured by a fully automated two-site TRACE immunoassay (BRAHMS Kryptor®, Brahms AG, Hennigsdorf, Germany) and TSH with a 3rd-generation CLIA assay (TSH-3, Advia Centaur, Bayer Corporation).

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of differentiated thyroid carcinoma
* total or near total thyroidectomy
* informed consent

Exclusion Criteria:

* no informed consent

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2003-09; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Martin Biermann, MD, Principal Investigator — Münster University Hospital
Locations (1):
- Department of Nuclear Medicine, Münster University Hospital, Münster, Germany

REFERENCES:
- [Result] Biermann M, Nofer JR, Riemann B, Lu J, Wilde J, Schober O. Clinical evaluation of a new highly sensitive thyroglobulin assay (Nichols Advantage®) in 99 patients with differentiated thyroid cancer (DTC) after total thyroidectomy [Abstract]. Clin Chem. 2004;50:A73.